CLINICAL TRIAL: NCT04049344
Title: Phase II Multicenter Open-Label Single-Arm Study of Decitabine Combined With Oxaliplatin in Patients With Relapsed/Metastatic Renal Cell Carcinoma
Brief Title: Decitabine Combined With Oxaliplatin in Patients With Advanced Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUCAS-025
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: renal cell carcinoma; chemotherapy; decitabine; oxaliplatin
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Decitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of decitabine with oxaliplatin treatment (Experimental): Patients receive Decitabine 10 mg/day for 5 consecutive days (d1-5) plus Oxaliplatin 75mg/m2 2-week-cycle (d6, d20) within 4 weeks. One cycle is defined as 4 weeks of treatment and total of 6 cycles are designed for patients.
  Interventions: Drug: Decitabine; Oxaliplatin

INTERVENTIONS:
Drug: Decitabine; Oxaliplatin — Patients receive Decitabine 10 mg/day for 5 consecutive days (d1-5) plus Oxaliplatin 75mg/m2 2-week-cycle (d6, d20) within 4 weeks. One cycle is defined as 4 weeks of treatment and total of 6 cycles are designed for patients.

SUMMARY:
The investigators reported previously that epigenetic activation of organic cation transporter (OCT2) by decitabine sensitizes RCC cells to oxaliplatin both in vitro and in xenografts. The objective of this phase II clinical trial is to investigate the efficacy and safety of sequential combination therapy with decitabine and oxaliplatin in patients with relapsed/metastatic renal cell carcinoma who progressed on standard of care.

DETAILED DESCRIPTION:
CHUCAS-025 (Cancer Hospital, University of Chinese Academy of Sciences) is a phase II trial conducted at 3 investigative centres in the Zhejiang Province, China. Eligible patients are 18 to 75 years old with relapsed/metastatic renal cell carcinoma progressed on standard of care. Patients receive Decitabine 10 mg/day for 5 consecutive days (d1-5) plus Oxaliplatin 75mg/m2 2-week-cycle (d6, d20) within 4 weeks. One cycle is defined as 4 weeks of treatment and total of 6 cycles are designed for patients. Patients who experienced unacceptable toxicities or clinical or documented progressive disease are discontinued from the study. The duration of any objective response is measured from the date the initial response is observed to the date that disease progression is observed. Patients receiving 2 cycles of treatment are considered evaluable for response using Response Evaluation Criteria in Solid Tumors (RECIST). Disease assessment by the investigator include response assessment and diagnostic imaging and measuring of target lesions. All patients receive computed tomography and/or magnetic resonance imaging scans for assessing disease status. All patients were followed up until death from any cause.

ELIGIBILITY:
Inclusion criteria

1. Age: 18 ~75 years old.
2. Patients who are diagnosed pathologically with relapsed/metastatic renal cell carcinoma have a disease progression on standard of care.
3. Performance status: Eastern Cooperative Oncology Group performance status ≦2.
4. Life expectancy more than 3 months.
5. Patients have adequate organ function, accord with following criteria: A. blood routine: Hemoglobin≥90g/L, absolute neutrophil count≥1.5×109/L, platelet count ≥ 80×109/L; B. Biochemical tests: total bilirubin is less than 1.5 times upper limit of normal, alanine aminotransferase and aspartate aminotransferase are less than 2.5 times upper limit of normal; C. creatinine less than 1.25 times upper limit of normal.
6. Patients agree to use adequate contraception in the period of trial and need negative pregnancy test in childbearing potential women.
7. Patients agree to receive treatment with epigenetic drugs.
8. Participant sign an institutional review board-approved, protocol-specific informed consent form in accordance with institutional guidelines.

Exclude criteria:

1. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
2. Organs failure.
3. ECOG >2.
4. Serious/active infection.
5. Autoimmune disorders or immunodeficiency diseases.
6. Patients with allergic constitution, or other disease need take drugs of immunosuppressant or corticosteroids.
7. Uncontrolled hypertension.
8. Myocardial ischemia (more than grade II ) or myocardial infarction or uncontrolled arrhythmia.
9. Cardiac insufficiency of grade III to IV according to NYHA criteria, or left ventricular ejection fraction (LVEF) <50%.
10. Coagulation disorders, tendency of haemorrhage, undergoing thrombolytic or anticoagulant therapy.
11. Unhealed wounds, or fractures.
12. With a history of psychotropic drug abuse or mental disorders.
13. Prior systemic therapies with any antitumor agents within 4 weeks.
14. With other uncurable cancers simultaneously.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Six months after randomization
  Progression free survival is defined as the time from randomization to first documented RECIST-defined tumor progression or death from any cause. Disease assessments are performed with the use of computed tomography or magnetic resonance imaging at baseline, every 8 weeks for the first year, and then every 12 weeks until disease progression or discontinuation of treatment. Imaging data were evaluated by the investigator to assess tumor response (according to RECIST version).

SECONDARY OUTCOMES:
Overall survival | Two years
  Overall survival is defined as the time from randomization to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Hua, Ph.D.; M.D., Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No